CLINICAL TRIAL: NCT01885910
Title: Use of Aczone 5% Gel as Maintenance Treatment of Acne Vulgaris Following Completion of Oral Doxycycline and Aczone 5% Gel Treatment
Brief Title: Aczone 5% Gel as Maintenance Treatment of Acne Vulgaris Following Completion of Oral Doxycycline and Aczone 5% Gel
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Derm Research, PLLC (Other)
Collaborators: WFH MEDICAL, LLC (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT-000508
Record Dates: First submitted 2013-06-21; First posted 2013-06-25 (Estimated); Results first posted 2015-02-26 (Estimated); Last update posted 2015-02-27 (Estimated); Status verified 2015-02

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — Doxycycline; Dapsone; Gels

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- doxy + aczone (Experimental): Subjects will start treatment with doxycycline 100mg once daily and Aczone 5% gel applied to the face twice daily and those who improve significantly are continued on Aczone gel alone to see if it can maintain therapeutic response
  Interventions: Drug: Doxycycline 100mg; Drug: Aczone 5% gel

INTERVENTIONS:
Drug: Doxycycline 100mg — Doxycycline 100mg by mouth once daily
  Other Names: Vibramycin, Oracea, Adoxa, Atridox
Drug: Aczone 5% gel — Aczone 5% gel twice daily
  Other Names: Dapsone

SUMMARY:
This pilot study will explore if continuation of treatment of treatment with Aczone 5% gel following combination treatment with with doxycycline and Aczone 5% gel can maintain therapeutic response.

DETAILED DESCRIPTION:
This is a two-center, open-label pilot study. The study is apprised of 7 study visits: Baseline and Weeks 4, 8, 12, 16, 20 and 24. All subjects will receive Aczone 5% gel BID and doxycycline 100mg by mouth once daily at Baseline. Those subjects achieving treatment response (i.e., IGA of 0, 1 or 2) at Week 12 will continue treatment with Aczone 5% gel BID at Week 12. Subjects not achieving treatment response will discontinue study participation.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient, male or female subjects of any race, age 12 or older. Female subjects of childbearing potential must have a negative urine pregnancy test result at Baseline and practice a reliable method of contraception throughout the study;
* Facial acne vulgaris characterized by the following:

IGA Score >3 10-50 facial inflammatory lesions (papules,pustules) 10-100 facial non-inflammatory lesions (open/closed comedones)

* Able to understand and comply with the requirements of the study and sign Informed Consent/HIPAA Authorization forms

Exclusion Criteria:

* Female subjects who are pregnant (positive urine pregnancy test), breast feeding, or who are of childbearing potential and not practicing a reliable method of birth control.
* Allergy/sensitivity to any component of the test treatment (Section 5.2), lincomycin, tetracyclines, or sulfites.
* Subjects who have not complied with the proper wash-out periods for prohibited medications/procedures (Supplement 1)>
* History of clinically significant anemia or hemolysis.
* History of enteritis (regional enteritis, ulcerative colitis, pseudomembranous colitis, or antibiotic-associated colitis).
* Skin disease/disorder that might interfere with the diagnosis or evaluation of acne vulgaris
* Evidence of recent alcohol or drug abuse
* Medical condition that, in the opinion of the Investigator, contraindicates the subject's participation in the clinical study
* History of poor cooperation, non-compliance with medical treatment or unreliability
* Participation in an investigational drug study within 30 days of the baseline visit.

Ages: 12 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2013-07; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leon H Kircik, MD, Principal Investigator — DermResearch, PLLC
Locations (1):
- DermResearch, PLLC, Louisville, Kentucky, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment at 2 sites for subjects at least 12 years of age with moderate to severe acne vulgaris began June 2013 and ended December 2013
Pre-assignment Details: Any subject might be excluded who is not at least 12 years of age, who does not have moderate to severe acne vulgaris based upon IGA score and lesion counts, who has not completed the proper washout of specified medications, or who has been in another investigational study 30 days prior
Groups:
- Doxy + Aczone: Subjects will start treatment with doxycycline 100mg once daily and Aczone 5% gel applied to the face twice daily
  Doxycycline 100mg and Aczone 5% gel: Subject is to take Doxycycline 100mg by mouth once daily and apply Aczone 5% gel to their face twice daily for 12 weeks; those subjects achieving treatment response will stop Doxycycline and continue applying Aczone 5% gel twice daily for 12 more weeks.
Period: Overall Study
Arm/Group | Doxy + Aczone
Started | 32
Completed | 24
Not Completed | 8

BASELINE CHARACTERISTICS:
Population: subjects at least 12 years of age who have moderate to severe acne vulgaris
Groups:
- Aczone/Doxy: subjects will take doxy 100mg daily and apply aczone 5% gel to the face twice daily for 12 weeks after which if their acne has improved they will continue on maintenance therapy of aczone gel for another 12 weeks
Arm/Group | Aczone/Doxy
Number analyzed (Participants) | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.8 (10.9)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 13
  Between 18 and 65 years | 19
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 12
Region of Enrollment [Number; unit: participants]
  United States | 32

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Remained Responders at Week 24
Description: At week 12 responder had an IGA <3 on a 6-point scale ranging from 0 (clear) to 5 (very severe) and at Week 24 this response was maintained
Time Frame: Assessed every 4 weeks, reported at Week 24
Population: only participants who were not lost to follow-up or did not withdraw consent were included in the final analysis
Measure: Number; unit: percentage of particpants
Arm/Group | Aczone/Doxy
Number analyzed (Participants) | 22
percentage of particpants | 82
Statistical Analysis 1: Comparison: Aczone/Doxy; Test type: Superiority or Other; p < .0001, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Inflammatory and Non-inflammatory Lesion Counts
Time Frame: Every 4 weeks
Population: participants with data
Measure: Mean (Standard Deviation); unit: lesions
Groups:
- Aczone/Doxy - Inflammatory: inflammatory lesion counts during treatment with aczone 5% and doxycycline 100mg
- Aczone/Doxy - Non Inflammatory: non inflammatory lesion counts during treatment with aczone 5% and doxy 100mg
Arm/Group | Aczone/Doxy - Inflammatory | Aczone/Doxy - Non Inflammatory
Number analyzed (Participants) | 31 | 31
lesions
  baseline | 27.3 (14.6) | 38.3 (20.8)
  week 16 (n=23,23) | 5.8 (4.9) | 10.0 (13.9)
  week 20 (n=23,23) | 7.3 (9.2) | 8.3 (11.6)
  week 24 (n=22,22) | 7.0 (9.1) | 6.6 (10.3)

3. Secondary Outcome: Percentage of Participants Who Are Responders at Week 16 and 20
Description: Responders is the percentage of participants who have an IGA <3 at Week 16 and 20
Time Frame: Assessed every 4 weeks, reported at weeks 16 and 20
Measure: Number; unit: percentage of participants
Arm/Group | Aczone/Doxy
Number analyzed (Participants) | 23
percentage of participants
  responders at week 16 | 78
  responders at week 20 | 87

4. Secondary Outcome: Nodule Counts
Description: number of nodules counted
Time Frame: every four weeks
Population: participants with data
Measure: Mean (Standard Deviation); unit: nodules
Arm/Group | Aczone/Doxy
Number analyzed (Participants) | 31
nodules
  Baseline | 0.4 (0.7)
  Week 16 (N=23) | 0.1 (0.4)
  Week 20 (N=23) | 0.1 (0.5)
  Week 24 (N=22) | 0.3 (0.9)

5. Secondary Outcome: Erythema
Description: the erythema severity scale ranges from 0 to 4 with 0 being no erythema and 4 being most extreme erythema
Time Frame: every 4 weeks
Population: participants with data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aczone/Doxy
Number analyzed (Participants) | 31
units on a scale
  Baseline | 1.3 (0.8)
  week 16 (N=23) | 0.7 (0.9)
  week 20 (N=23) | 0.9 (0.8)
  week 24 (N=22) | 1.1 (0.9)

6. Secondary Outcome: Dryness
Description: the dryness severity scale ranges from 0 to 4 with 0 being no dryness and 4 being most extreme dryness
Time Frame: every 4 weeks
Population: participants with data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aczone/Doxy
Number analyzed (Participants) | 31
units on a scale
  baseline | 0.6 (0.8)
  week 16 (N=23) | 0.3 (0.6)
  week 20 (N=23) | 0.1 (0.3)
  week 24 (N=22) | 0.1 (0.3)

7. Secondary Outcome: Peeling
Description: the peeling severity scale ranges from 0 to 4 with 0 being no peeling and 4 being most extreme peeling
Time Frame: every four weeks
Population: participants with data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aczone/Doxy
Number analyzed (Participants) | 31
units on a scale
  baseline | 0.4 (0.9)
  week 16 (N=23) | 0.1 (0.3)
  week 20 (N=23) | 0.1 (0.3)
  week 24 (N=22) | 0.1 (0.3)

8. Secondary Outcome: Oiliness
Description: the oiliness severity scale ranges from 0 to 10 with 0 being no oiliness and 10 being most extreme oiliness
Time Frame: every 4 weeks
Population: participants with data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aczone/Doxy
Number analyzed (Participants) | 31
units on a scale
  baseline | 1.6 (1.1)
  week 16 (N=23) | 0.8 (0.8)
  week 20 (N=23) | 0.6 (0.7)
  week 24 (N=22) | 0.3 (0.5)

9. Secondary Outcome: Pruritis
Description: the pruritis severity scale ranges from 0 to 5 with 0 being no pruritis and 5 being the most extreme pruritis
Time Frame: every 4 weeks
Population: participants with data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aczone/Doxy
Number analyzed (Participants) | 31
units on a scale
  baseline | 0.4 (0.8)
  week 16 (N=23) | 0.2 (0.6)
  week 20 (N=23) | 0.1 (0.3)
  week 24 (N=22) | 0 (0.2)

10. Secondary Outcome: Burning
Description: the burning severity scale ranges from 0 to 10 with 0 being no burning and 10 being most extreme burning
Time Frame: every 4 weeks
Population: participants with data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aczone/Doxy
Number analyzed (Participants) | 31
units on a scale
  baseline | 0.1 (0.5)
  week 16 (N=23) | 0.1 (0.4)
  week 20 (N=23) | 0 (0)
  week 24 (N=22) | 0 (0.2)

ADVERSE EVENTS:
Time Frame: 6 months
Description: Subjects were interviewed regarding changes in their health and the severity of pruritis and burning at each study visit; each subject was graded at each study visit regarding their current severity of erythema, dryness, peeling and oiliness on a 5-point scale.
Arm/Group | Doxy + Aczone
Serious Adverse Events (participants affected / at risk) | 0/32
Other Adverse Events (participants affected / at risk) | 7/32
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Doxy + Aczone (N=32)
nausea (Gastrointestinal disorders) | 3 (3) — resolved, no residual effects
burning (Skin and subcutaneous tissue disorders) | 1 (1) — not resolved, f/u deemed unnecessary
vomiting (Gastrointestinal disorders) | 1 (1) — resolved, no residual effects
headache (Vascular disorders) | 1 (1) — resolved, no residual effects
pruritis (Skin and subcutaneous tissue disorders) | 1 (1) — resolved, no residual effects

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes